CLINICAL TRIAL: NCT01534819
Title: Aneurysm Treatment Using the Heli-FX™ EndoAnchor™ System Global Registry
Brief Title: ANCHOR (Aneurysm Treatment Using the Heli-FX™ EndoAnchor™ System Global Registry)
Acronym: ANCHOR
Status: Active, not recruiting | Type: Observational
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: Anchor Post Market Registry
Record Dates: First submitted 2012-02-09; First posted 2012-02-17 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Aortic Aneurysm
Keywords: Endograft; Endurant; Heli-FX™; EndoAnchor™; Short neck; Endovascular treatment; Interventional treatment of aortic aneurysm; Abdominal aortic aneurysm; AAA; Thoracic aortic aneurysm; TAA; Advanced disease
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Abdominal; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Protocol B, abdominal arm, revision group: AAA subjects with previously implanted commercial endografts for the treatment of graft migration and/or Type Ia endoleak
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament
- Protocol B, abdominal arm, primary group: AAA subjects at the time of initial endograft implantation either to prevent endograft migration and Type Ia endoleak, or to treat Type Ia endoleak evident at the time of implantation.
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament
- Protocol B, thoracic arm, revision group: TAA subjects with previously implanted commercial endografts for the treatment of migration and/or Type Ia and/or Type Ib endoleak at the proximal or distal attachment site
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament
- Protocol B, thoracic arm, primary group: TAA subjects at the time of initial endograft implantation either to prevent endograft migration and Type I endoleak, or to treat Type Ia and/or Ib endoleak at the proximal or distal attachment site evident at the time of implantation
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament
- Protocol B, advanced disease arm, revision group: Advanced disease subjects with previously implanted commercial endografts for the treatment of migration and/or Type Ia and/or Type Ib endoleak at the proximal or distal attachment site
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament
- Protocol B, advanced disease arm, primary group: Advanced disease subjects at the time of initial endograft implantation either to prevent endograft migration and Type I endoleak, or to treat Type Ia and/or Ib endoleak at the proximal or distal attachment site evident at the time of implantation.
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament
- Protocol C, abdominal arm, short neck, primary group: Planned use of Heli-FX™ in conjunction with the Endurant II/IIs endograft in AAA subjects with short proximal necks (≥ 4 mm and < 10 mm) in primary group.
  Interventions: Device: EndoAnchor™; Procedure: endovascular treament

INTERVENTIONS:
Device: EndoAnchor™ — Use of the EndoAnchor™ in conjunction with endograft
  Other Names: Heli-FX™; Heli-FX™ EndoAnchor™ System
Procedure: endovascular treament — implantation of a device inserted through an artery

SUMMARY:
The ANCHOR registry is a multi-center, post-market, non-interventional, non-randomized, prospective study.

Subjects must sign an ICF prior to obtaining any study specific information. Subjects are eligible to be consented up to 30 days post-procedure.

Enrolled subjects will be followed as per local 'standard of care' for up to 5 years post procedure. Study recommended follow-up is per SVS and ESVS guidance.

DETAILED DESCRIPTION:
The objective of the ANCHOR registry is to expand the clinical knowledge based on the use of the Heli-FX™ EndoAnchor™ System. This registry will include "real world" use over a broad spectrum of geographies, by a wide variety of practicing clinicians, and with a minimal degree of subject selection criteria.

ELIGIBILITY:
Protocol B:

Inclusion criteria:

1. Subjects with asymptomatic, symptomatic, or ruptured aortic aneurysms
2. Subject ≥ 18 years old
3. Subject has provided written informed consent, either before or less than or equal to 30 calendar days after the index procedure
4. Subject is willing and able to comply with standard of care followup evaluations
5. Subject has a previously implanted endograft or will be undergoing repair, with one of the following aortic aneurysm endograft devices:

   * Cook Zenith or Cook Zenith TX2
   * Gore Excluder or TAG
   * Medtronic AneuRx
   * Medtronic Talent
   * Medtronic Endurant or Valiant
   * Any additional third party AAA endograft device that is commercially available and listed as compatible with Heli-FX™ in the IFU
6. Subject's iliac/femoral access is compatible with:

   * a 16 French sheath (abdominal subjects)
   * 18 French sheath (thoracic subjects)
   * Selected 16 or 18 French sheath, as applicable to the device selected for use (advanced disease subjects)
7. Subject has a previously implanted endograft that has migrated or has a Type I endoleak within the aorta or will undergo implantation of an endograft that in the opinion of the investigator will be at increased risk of such complications

Exclusion criteria:

1. Subject has known allergy to the EndoAnchor™ implant material (nickel, chromium, molybdenum, or cobalt)
2. Subject has a life expectancy of less than 1 year
3. Subject is participating in a clinical study or registry that, in the Investigator's opinion, may conflict or may have a negative impact on the subject's safety
4. Subject was treated with EndoAnchor™ in the same segment of the aorta that will be treated in the registry
5. Subject has an active or known history of bleeding diathesis
6. Subject has a condition that threatens to infect the endograft (active bacteremia, or infections that carry increased risk of endograft infection)
7. Significant thrombus or calcium at the location of planned EndoAnchor™ implantation that precludes adequate EndoAnchor™ penetration of the aortic wall
8. Use where, for whatever reason, each EndoAnchor™ is not anticipated to adequately penetrate into the aortic wall
9. Subject has an aortic dissection that involves an area to be treated with EndoAnchor™
10. Subject has Marfan Syndrome, Ehlers Danlos Syndrome, or another collagen vascular disease
11. Subject is pregnant

Protocol C:

Inclusion criteria:

* Subjects with asymptomatic or symptomatic abdominal aortic aneurysms that will receive the Heli-FX™ in conjunction with the Endurant II/IIs endograft as part of their planned EVAR treatment
* Subject ≥ 18 years old
* Subject has provided written informed consent, either before or less than or equal to 30 calendar days after the index procedure
* Subject is willing and able to comply with standard of care followup evaluations
* Subject will be undergoing AAA repair with the bifurcated main body Endurant II/IIs stent graft in conjunction with Heli-FX™ with a proximal neck length of ≥ 4mm to < 10mm and treated in accordance with the Endurant II/IIs and Heli-FX™ IFUs
* Subject's iliac/femoral access is compatible with a 16 French sheath

Exclusion criteria:

* Subject has known allergy to the EndoAnchor™ implant material (nickel, chromium, molybdenum, or cobalt)
* Subject has a life expectancy of less than 1 year
* Subject is participating in a clinical study or registry that, in the Investigator's opinion, may conflict or may have a negative impact on the subject's safety
* Subject was previously treated with EndoAnchor™ implants in the same segment of the aorta that will be treated within the registry, or has a previously implanted AAA endograft that has migrated or has a Type Ia endoleak, or is being treated for a ruptured abdominal aortic aneurysm, or has planned usage of an Endurant II/IIs AUI main body stent graft configuration
* Subject has an active or known history of bleeding diathesis
* Subject has a condition that threatens to infect the endograft (active bacteremia, or infections that carry increased risk of endograft infection)
* Significant thrombus or calcium at the location of planned EndoAnchor™ device implantation that precludes adequate EndoAnchor™ implant penetration of the aortic wall
* Use where, for whatever reason, each EndoAnchor™ implant is not anticipated to adequately penetrate into the aortic wall
* Subject has an aortic dissection that involves an area to be treated with EndoAnchor™ implants
* Subject has Marfan Syndrome, Ehlers Danlos Syndrome, or another collagen vascular disease
* Subject is pregnant
* Physician does not intend to treat subject on-label per the Endurant II/IIs and Heli-FX™ IFU requirements or if the physician intends to use Heli-FX™ in a chimney procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Protocol B: subjects with AAA, TAA, or advanced aortic aneurysmal disease treated with the Heli-FX™ EndoAnchor™ System in conjunction with commercially available abdominal and thoracic Endografts, in both "Primary" and "Revision" settings and who meet the inclusion/exclusion criteria.
  Protocol C:The intended population will include those subjects with short (≥ 4 mm and < 10 mm) infrarenal proximal neck lengths who are appropriate candidates for infrarenal AAA treatment with the Heli-FX™ EndoAnchor™ System in conjunction with the Endurant II/IIs endograft system and who meet the inclusion/exclusion criteria
Sampling Method: Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2026-04-24 (Estimated)

PRIMARY OUTCOMES:
Protocol B has composite primary safety endpoints, tabulated separately for the abdominal, thoracic and advanced disease arms | Through 12 months
  The primary safety endpoint is defined by:
  i. freedom from device-related serious adverse events at 12 months and ii. freedom from procedure-related serious adverse events at 12 months iii. freedom from aneurysm-related mortality defined as: i. death within 30 days of the index procedure ii. death within 30 days of a secondary procedure to address the aneurysm iii. death from rupture of the treated aneurysm
Protocol B has composite primary effectiveness endpoints, tabulated separately for the abdominal, thoracic and advanced disease arms | Through 12 months
  The primary effectiveness endpoint requires all of the following:
  i successful implantation of the minimum number of EndoAnchor™ and ii freedom from migration at 12 months and iii freedom from Type I endoleak at the targeted attachment site(s) at 12 months
Protocol C has composite primary safety endpoint | Through 12 months
  The primary safety endpoint is defined by:
  1. device-related serious adverse events at 12 months
  2. aneurysm-related mortality defined as:
  i. death within 30 days of the index procedure ii. death within 30 days of a secondary procedure to address the aneurysm iii. death from rupture of the treated aneurysm
Protocol C have composite primary effectiveness endpoint | Through 12 months
  The primary effectiveness endpoint is treatment success which is defined as the successful implantation of EndoAnchor™ implants at the index procedure, and the absence of:
  1. migration at 12 months and
  2. Type I endoleak at the targeted attachment site(s) at 12 months

SECONDARY OUTCOMES:
Protocol B has the secondary endpoints chosen to reflect the clinical success and safety of Heli-FX™. Each of the secondary endpoints will be measured individually at 30 days and 12 months and yearly thereafter. | Through 5 years
  1. Technical success defined as successful deployment of EndoAnchor™ at their intended location. Technical success will be assessed separately for the target attachment sites; proximally and/or distally
  2. Clinical success will be defined as the successful implantation of the suggested number of EndoAnchor™ at the index procedure, and the absence of: death as a result of aneurysm-related treatment; Type Ia endoleak; Type Ib endoleak (TAA and advanced disease only); endograft infection; endograft migration; loss of endograft fabric integrity as a result of the EndoAnchor™; Rupture of the treated aneurysm; Conversion to open surgical repair
  3. Secondary aneurysm-related interventions after EndoAnchor™ implantation
  4. all-cause mortality
  5. Freedom from EndoAnchor™ fracture
Protocol C has the secondary endpoints chosen to reflect the clinical success and safety of Heli-FX™. Each of the secondary endpoints will be measured individually at 30 days and 12 months and yearly thereafter. | Through 5 years
  1. Technical success defined as successful deployment of EndoAnchor™ at their intended location. Technical success will be assessed separately for the target attachment sites; proximally and/or distally
  2. Clinical success will be defined as the successful implantation of EndoAnchor™ at the index procedure, and the absence of: aneurysm-related mortality; Type Ia endoleak; endograft infection; endograft migration; loss of endograft fabric integrity as a result of the EndoAnchor™; Rupture of the treated aneurysm; Conversion to open surgical repair
  3. Secondary aneurysm-related interventions after EndoAnchor™ implantation
  4. all-cause mortality
  5. EndoAnchor™ implant fracture

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul de Vries, MD, Principal Investigator — Universitair Medisch Centrum Groningen, Netherlands; William Jordan, MD, Principal Investigator — Augusta University Health, United States
Locations (87):
- United States (46):
  - University of Alabama, Birmingham, Alabama
  - Abrazo Arizona Heart Institute, Phoenix, Arizona
  - John L McClellan Memorial Veterans Hospital, Little Rock, Arkansas
  - VA Loma Linda Medical Center, Loma Linda, California
  - El Camino Hospital, Mountain View, California
  - University of California Irvine Medical Center, Torrance, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital Vascular Surgery Dept., Washington D.C., District of Columbia
  - Baptist Cardiac & Vascular Institute, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Kaiser Permanente Moanalua Medical Center and Clinic, Honolulu, Hawaii
  - HeartCare Midwest, Peoria, Illinois
  - Evanston Hospital, Skokie, Illinois
  - Southern Illinois University, Springfield, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess-Harvard, Boston, Massachusetts
  - Michigan Vascular Center, Flint, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Washington University School of Medicine, Barnes Jewish West County Hospital, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Albany Medical Center, Albany, New York
  - New York University Langone Medical Center, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Maimonides Medical Center, New York, New York
  - Vascular Health Partners, Queensbury, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - University of North Carolina (UNC) Memorial Hospital, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Pinnacle Harrisburg Campus, Wormleysburg, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - CHI Memorial Hospital Chattanooga, Chattanooga, Tennessee
  - Baptist Memorial Hospital-Memphis, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Scott and White Medical Center, Temple, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Harborview Medical Center, University of Washington, Seattle, Washington
- Australia (5):
  - Concord Repatriation General Hospital, Concord
  - Dandenong Hospital, Dandenong
  - Royal Perth Hospital, Perth
  - Sir Charles Gairdner Hospital, Perth
  - Royal North Shore Hospital, St Leonards
- Austria (2):
  - A.ö. Landeskrankenhaus - Universitätskliniken Innsbruck, Innsbruck
  - Allgemeines Krankenhaus - Universitätskliniken Wien, Vienna
- France (2):
  - Hôpital Pontchaillou, Rennes
  - Nouvel Hôpital Civil, Strasbourg
- Germany (10):
  - Medizinische Fakultät der RWTH, Aachen
  - Deutsches Herzzentrum, Berlin
  - University Hospital Heidelberg, Heidelberg
  - Park Hospital Leipzig, Leipzig
  - St. Bonifatius Hospital, Lingen
  - Klinikum Ludwigsburg, Ludwigsburg
  - LMU Kilinikum der Universitaet Muenchen, Munich
  - Technical University of Munich, Munich
  - St. Franzsikus-Hospital GmbH, Münster
  - Klinikum Nuremberg, Nuremberg
- Italy (5):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - AO Universitaria Policlinico, Roma
  - Unihospital San Giovanni di Dio Ruggi d'Aragona, Salerno
  - University of Siena, Siena
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Torino
- Netherlands (5):
  - Rijnstate Hospital, Arnhem
  - Medisch Spectrum Twente, Enschede
  - St. Antonius Hospital, Nieuwegein
  - Maasstad Hospital Rotterdam, Rotterdam
  - UMC Utrecht, Utrecht
- Auckland City Hospital, Auckland, New Zealand
- Narodny ustav srdcovych a cievnych chorob, Nové Mesto, Slovakia
- Spain (3):
  - Thorax Institute Hospital Clinic, Barcelona
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Hospital Clínico Universitario de Valladolid, Valladolid
- Malmo University Hospital, Malmo, Sweden
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitätsSpital Zürich, Zurich
- United Kingdom (4):
  - The Royal Liverpool and NHS Broadgreen University Hospitals - Royal Liverpool University Hospital, Liverpool
  - Imperial College Healthcare NHS Trust, London
  - Wythenshawe Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jordan WD Jr, Mehta M, Varnagy D, Moore WM Jr, Arko FR, Joye J, Ouriel K, de Vries JP; Aneurysm Treatment using the Heli-FX Aortic Securement System Global Registry (ANCHOR) Workgroup Members. Results of the ANCHOR prospective, multicenter registry of EndoAnchors for type Ia endoleaks and endograft migration in patients with challenging anatomy. J Vasc Surg. 2014 Oct;60(4):885-92.e2. doi: 10.1016/j.jvs.2014.04.063. Epub 2014 Jul 31. PMID 25088739
- [Result] Jordan WD Jr, Mehta M, Ouriel K, Arko FR, Varnagy D, Joye J, Moore WM Jr, de Vries JP. One-year results of the ANCHOR trial of EndoAnchors for the prevention and treatment of aortic neck complications after endovascular aneurysm repair. Vascular. 2016 Apr;24(2):177-86. doi: 10.1177/1708538115590727. Epub 2015 Jun 10. PMID 26069087
- [Derived] Arko FR 3rd, Pearce BJ, Henretta JP, Fugate MW, Torsello G, Panneton JM, Peng Y, Edward Garrett H Jr. Five-year outcomes of endosuture aneurysm repair in patients with short neck abdominal aortic aneurysm from the ANCHOR registry. J Vasc Surg. 2023 Dec;78(6):1418-1425.e1. doi: 10.1016/j.jvs.2023.07.058. Epub 2023 Aug 7. PMID 37558144
- [Derived] van Noort K, Vermeulen JJM, Goudeketting SR, Ouriel K, Jordan WD Jr, Panneton JM, Slump CH, de Vries JPM. Sustainability of Individual EndoAnchor Implants in Therapeutic Use to Treat Type Ia Endoleak After Endovascular Aneurysm Repair. J Endovasc Ther. 2019 Jun;26(3):369-377. doi: 10.1177/1526602819837753. Epub 2019 Mar 25. PMID 30907259
- [Derived] Arko FR 3rd, Stanley GA, Pearce BJ, Henretta JP, Fugate MW, Mehta M, Torsello G, Panneton JM, Garrett HE Jr. Endosuture aneurysm repair in patients treated with Endurant II/IIs in conjunction with Heli-FX EndoAnchor implants for short-neck abdominal aortic aneurysm. J Vasc Surg. 2019 Sep;70(3):732-740. doi: 10.1016/j.jvs.2018.11.033. Epub 2019 Mar 6. PMID 30850297
- [Derived] Muhs BE, Jordan W, Ouriel K, Rajaee S, de Vries JP. Matched cohort comparison of endovascular abdominal aortic aneurysm repair with and without EndoAnchors. J Vasc Surg. 2018 Jun;67(6):1699-1707. doi: 10.1016/j.jvs.2017.10.059. Epub 2017 Dec 18. PMID 29248241
- [Derived] Jordan WD Jr, de Vries JP, Ouriel K, Mehta M, Varnagy D, Moore WM Jr, Arko FR, Joye J, Henretta J. Midterm outcome of EndoAnchors for the prevention of endoleak and stent-graft migration in patients with challenging proximal aortic neck anatomy. J Endovasc Ther. 2015 Apr;22(2):163-70. doi: 10.1177/1526602815574685. PMID 25809354
- [Derived] Jordan WD Jr, Ouriel K, Mehta M, Varnagy D, Moore WM Jr, Arko FR, Joye J, de Vries JP; Aneurysm Treatment using the Heli-FX Aortic Securement System Global Registry ANCHOR; Aneurysm Treatment using the Heli-FX Aortic Securement System Global Registry ANCHOR. Outcome-based anatomic criteria for defining the hostile aortic neck. J Vasc Surg. 2015 Jun;61(6):1383-90.e1. doi: 10.1016/j.jvs.2014.12.063. Epub 2015 Feb 28. PMID 25735260
- [Derived] de Vries JP, Ouriel K, Mehta M, Varnagy D, Moore WM Jr, Arko FR, Joye J, Jordan WD Jr; Aneurysm Treatment Using the Heli-FX Aortic Securement System Global Registry ANCHOR Trial. Analysis of EndoAnchors for endovascular aneurysm repair by indications for use. J Vasc Surg. 2014 Dec;60(6):1460-7.e1. doi: 10.1016/j.jvs.2014.08.089. Epub 2014 Oct 3. PMID 25284629
- See also: Medtronic — http://www.medtronic.com